CLINICAL TRIAL: NCT04347226
Title: A Randomized Phase 2 Study of Anti-IL-8 Therapy Versus Standard of Care in the Treatment of Hospitalized Patients With Severe COVID-19
Brief Title: Anti-Interleukin-8 (Anti-IL-8) for Patients With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis indicated that futility boundary was reached.
Sponsor: Columbia University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Mark Stein, Associate Professor of Medicine at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS9881
Record Dates: First submitted 2020-04-02; First posted 2020-04-15 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor; Sars-CoV2; Hematological Malignancy
Keywords: COVID-19; coronavirus; corona virus; COVID
MeSH Terms: conditions — Hematologic Neoplasms; COVID-19; Coronavirus Infections | interventions — HuMax-IL8

STUDY DESIGN:
Intervention Model Description: Participants will receive either BMS-986253 2400mg intravenous (IV) at 0 and 2 weeks (if patient is still hospitalized) and then 4 weeks (only if continued severe respiratory disease) or standard of care treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986253 (Experimental): BMS-986253 2400mg IV
  Interventions: Drug: BMS-986253
- Standard of Care treatment (No Intervention): Usual treatment of COVID-19 per study physician discretion

INTERVENTIONS:
Drug: BMS-986253 — BMS-986253 2400mg IV at 0 and 2 weeks (if patient is still hospitalized) and then 4 weeks (only if still hospitalized with continued severe respiratory disease).
  Arms: BMS-986253

SUMMARY:
This study is for patients that are hospitalized for Coronavirus Disease 2019 (COVID-19). The purpose of this study is to see whether neutralizing interleukin-8 (IL-8) with BMS-986253 can help improve the health condition of participants infected with COVID-19. This is the first in-human study of this investigational product specifically in patients with severe COVID-19. Currently there are no FDA approved medications that improve the chance of survival in patients diagnosed with COVID-19. However there are usual treatments currently being used to help treat COVID-19 patients and BMS-986253 will be compared to these standard of care treatments in this study.

DETAILED DESCRIPTION:
This is a single center, randomized, open-label, phase 2 trial to evaluate the time-to-improvement in the 7 point ordinal scale following treatment with anti-IL-8 therapy (BMS-986253) compared to standard of care in hospitalized patients with COVID-19 respiratory disease. Patients will be randomized 2:1 to receive either BMS-986253 or standard of care. Patients randomized to treatment with BMS-986253 will receive between 1-3 doses of therapy depending on their clinical status. Participants will be assessed daily while in the hospital and with then be followed for up to 1 year after discharge.

ELIGIBILITY:
Inclusion Criteria

* Male or female adult ≥ 18 years of age at time of enrollment.
* Confirmed diagnosis of SARS-CoV-2 infection ≤ 14 days prior to registration.
* Inpatient hospitalization (or documentation of a plan to admit to the hospital if the patient is in the emergency department)
* Evidence of pneumonia by chest radiographs, chest CT OR chest auscultation (rales, crackles).
* Severe respiratory disease (oxygen saturation ≤93% on room air and requiring supplemental oxygen) OR critical respiratory disease (requiring non-rebreather, non-mechanical/mechanical ventilation, high-flow nasal cannula, ICU admission).
* Patients can continue their anti-cancer therapy at the discretion of the treating physician.
* Adequate laboratory tests including:

  * absolute neutrophil count (ANC) >500 cells/mm3
  * Platelet count >20,000 cells/mm3
  * Serum total bilirubin <1.5 × upper limit of normal (ULN)
  * alanine aminotransferase (ALT) <5 × ULN
  * aspartate aminotransferase (AST) <5 × ULN
* Age and Reproductive Status

  1. Males and females, aged at least 18 years old
  2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study treatment.
  3. Women must not be breastfeeding.
  4. WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment plus for a total of 155 days post treatment completion. Local laws and regulations may require use of alternative and/or additional contraception methods.
  5. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, but should still undergo pregnancy testing as described in this section.
  6. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception during study treatment with BMS-986253 for a total of 215 days post-treatment completion.
  7. Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, and still must undergo pregnancy testing as described in this section.
* Willingness to provide written informed consent and HIPAA authorization for the release of personal health information, and the ability to comply with the study requirements (note: HIPAA authorization will be included in the informed consent). In cases of partial impairment, impairment that fluctuates over time, or complete impairment due to dementia, stroke, traumatic brain injury, developmental disorders (including mentally disabled persons), serious mental illness, delirium, medical sedation, or intubation, a subject may be enrolled if the subject's legally authorized representative consents on the subject's behalf.

Exclusion Criteria

* Treatment with anti-IL-6, anti-IL-6R antagonists or Janus kinase inhibitor (JAKi) within 48 hours of first dose of study treatment.
* No other investigational therapies with the intent to treat the patient's COVID-19 can be administered while the patient is enrolled in the study.

  o Exception is remdesivir, hydroxychloroquine or other treatments being used as compassionate use for COVID-19.
* Expected non-COVID-related survival of < 2 months.
* Ongoing systemic immunosuppressive therapy ≤ 14 days prior to study treatment administration (except for adrenal replacement steroid doses ≤ 10mg daily prednisone equivalent in the absence of active autoimmune disease or a short course of steroids (<5 days) up to 7 days prior to initiating study treatment).
* Receipt of non-oncology vaccines containing live virus for prevention of infectious diseases within 4 weeks prior to first dose of study treatment
* History of severe hypersensitivity reaction to any monoclonal antibody (mAb)
* Multi-organ failure requiring vasopressors or continuous veno-venous hemofiltration (CVVH) or extracorporeal membrane oxygenation.
* No active systemic bacterial or fungal infection o Patients with a history of positive bacterial or fungal cultures but on enrollment do not have suspected or known active systemic bacterial or fungal infections are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark N Stein, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BMS-986253 | Standard of Care Treatment
Started | 29 | 14
Completed | 29 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986253 | Standard of Care Treatment | Total
Number analyzed (Participants) | 29 | 14 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (13.1) | 73.0 (10.9) | 69.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 15 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 7 | 20
  Not Hispanic or Latino | 16 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 8 | 4 | 12
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 8 | 5 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 14 | 43

OUTCOME MEASURES:

1. Primary Outcome: Time to Improvement in the 7-point Ordinal Scale
Description: The time to improvement in the 7-point ordinal scale in patients treated with anti-IL-8 therapy compared to standard of care/controls. Measured from baseline to 2 point or greater improvement in 7-point ordinal scale.
Time Frame: Up to 10.5 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BMS-986253 | Standard of Care Treatment
Number analyzed (Participants) | 29 | 14
days | 12 [5 to 57] | 6 [4 to 13]

2. Secondary Outcome: Time to Death
Description: The time to death will be defined as the time from onset from symptoms until death from any cause. Patients who are alive or lost to follow-up at the cut-off date will be censored from this analysis.
Time Frame: Up to 10.5 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BMS-986253 | Standard of Care Treatment
Number analyzed (Participants) | 29 | 14
days | 30 [15 to NA] — upper limit of 95% Confidence Interval not reached due to insufficient number of participants with events | NA [14 to NA] — median and upper limit of 95% Confidence Interval not reached due to insufficient number of participants with events

3. Secondary Outcome: Time to Intubation
Description: The time to intubation will be defined as the time from symptom onset until time of intubation. Any patients already intubated at enrollment will be censored from this analysis.
Time Frame: Up to 10.5 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | BMS-986253 | Standard of Care Treatment
Number analyzed (Participants) | 29 | 14
days | 11.5 [10.2 to 14.2] | 3 [3 to 3]

4. Secondary Outcome: Proportion of Patients Requiring ICU Admission
Description: The proportion of patients requiring intensive care unit (ICU) admission will be calculated as the number of patients requiring ICU admission over the course of their hospitalization over the number of evaluable patients.
Time Frame: Up to 10.5 months
Measure: Number; unit: participants
Arm/Group | BMS-986253 | Standard of Care Treatment
Number analyzed (Participants) | 18 | 4
participants | 9 | 1

5. Secondary Outcome: Mortality at 1 Month
Description: Number of participants who have died 1 month from the time of start of treatment
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986253 | Standard of Care Treatment
Number analyzed (Participants) | 29 | 14
Participants | 8 | 4

ADVERSE EVENTS:
Time Frame: Up to 10.5 months
Arm/Group | BMS-986253 | Standard of Care Treatment
All-Cause Mortality (participants affected / at risk) | 11/29 | 5/14
Serious Adverse Events (participants affected / at risk) | 11/29 | 4/14
Other Adverse Events (participants affected / at risk) | 20/29 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS-986253 (N=29) | Standard of Care Treatment (N=14)
Infections and infestation (Infections and infestations) | 5 (5) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS-986253 (N=29) | Standard of Care Treatment (N=14)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 2 (9) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (7) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (11) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Infections and infestations (Infections and infestations) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (5) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
International Normalised Ratio (INR) (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT04347226/Prot_SAP_000.pdf